CLINICAL TRIAL: NCT01079520
Title: A Prospective Trial of Endobronchial Ultrasound- Transbronchial Needle Aspiration Compared to Mediastinoscopy for Mediastinal Lymph Node Staging of Non-small Cell Lung Cancer
Brief Title: Endobronchial Ultrasound- Transbronchial Needle Aspiration (EBUS-TBNA) Versus Mediastinoscopy for Mediastinal Lymph Node Staging of Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sang-Won Um, Assistant Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-08-053; CRS110-19-1 (Other Grant/Funding Number: Samsung Medical Center Clinical Research Development Program)
Record Dates: First submitted 2010-01-20; First posted 2010-03-03 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Cancer; Lung Cancer; Ultrasound; Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms | interventions — Mediastinoscopy

INTERVENTIONS:
Procedure: Endobronchial ultrasound (EBUS) — Minimally invasive technique to stage lung cancers
Procedure: Mediastinoscopy — Traditional surgical method to stage lung cancers

SUMMARY:
Accurate staging of the mediastinum is essential to evaluate prognosis in non-small cell lung cancer and to devise an appropriate treatment plan. Mediastinal staging by surgical techniques (mainly cervical mediastinoscopy) is considered to be the gold standard, although surgical staging is invasive, requires general anesthesia, and is subject to potential serious complications. Endobronchial ultrasound (EBUS)-transbronchial needle aspiration (TBNA) is a new modality for the evaluation of mediastinal and hilar lymph node metastasis from lung cancer. Compared to other diagnostic methods, EBUS-TBNA is a real-time procedure that enables multiple biopsies with high-quality histologic cores under local anesthesia. However, there have been few data on the head-to-head comparisons of mediastinoscopy and EBUS-TBNA. The aim of this prospective study is to determine the sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of EBUS-TBNA and mediastinoscopy in identifying N2 and N3 lymph node for patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histology-proven non-small cell lung cancer
* N2 or N3 lymph node invasion is suspected based on chest CT or PET/CT scans (at least one of three criteria) : 1) enlarged (1cm or more in short axis diameter) mediastinal lymph node(s), 2) FDG uptake in the mediastinal lymph node(s), or 3) FDG uptake in N1 node(s)
* The patient is otherwise considered a candidate for a surgical treatment with the intention to cure

Exclusion Criteria:

* Distant metastasis
* Inoperable T4 disease
* Confirmed supraclavicular lymph node metastasis
* Former therapy (chemotherapy or radiotherapy or surgery) for lung cancer
* Contraindications for bronchoscopy
* Uncorrected coagulopathy
* Concurrent other malignancies
* Suspicious mediastinal lymph node metastasis which are not accessible by EBUS-TBNA or mediastinoscopy (i.e. paraaortic, aortopulmonary window, or paraesophageal lymph nodes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of the study is to compare the sensitivity of EBUS-TBNA vs. mediastinoscopy. | 1 month interval

SECONDARY OUTCOMES:
The secondary outcome measures of the study are to compare the specificity, negative predictive value, positive predictive value, and accuracy of EBUS-TBNA vs. mediastinoscopy. | 1 month interval

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Won Um, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Um SW, Kim HK, Jung SH, Han J, Lee KJ, Park HY, Choi YS, Shim YM, Ahn MJ, Park K, Ahn YC, Choi JY, Lee KS, Suh GY, Chung MP, Kwon OJ, Kim J, Kim H. Endobronchial ultrasound versus mediastinoscopy for mediastinal nodal staging of non-small-cell lung cancer. J Thorac Oncol. 2015 Feb;10(2):331-7. doi: 10.1097/JTO.0000000000000388. PMID 25611227